CLINICAL TRIAL: NCT05378425
Title: A Phase 1, First-in-Human Study of NTX-1088, a Monoclonal Antibody Targeting the Poliovirus Receptor (PVR, CD155), as Monotherapy and Combined With Pembrolizumab, in Patients With Advanced Solid Malignancies
Brief Title: A Study of NTX-1088, a Monoclonal Antibody Targeting the Poliovirus Receptor (PVR, CD155), as Monotherapy and Combined With Pembrolizumab
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nectin Therapeutics Ltd (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NTX 1088-01; KEYNOTE-E92 (Other: Merck Sharp & Dohme, LLC); MK-3475-E92 (Other: Merck Sharp & Dohme, LLC)
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Tumor, Solid; Advanced Solid Tumor; Metastatic Cancer; Locally Advanced Solid Tumor
Keywords: PVR; IO; Immune Oncology
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 - Dose Escalation Phase (Monotherapy) (Experimental): NTX-1088 administered as a 60-minute IV infusion at escalating doses as a monotherapy. NTX-1088 will be administered on Day 1 of a 21-day cycle.
  Interventions: Drug: NTX-1088
- Part 1 - Dose Escalation Phase (Combination Therapy) (Experimental): NTX-1088 administered as a 60-minute IV infusion in escalating doses in combination with pembrolizumab. NTX-1088 will be administered on Day 1 of a 21-day cycle.
  Pembrolizumab will be administered as a 30-minute IV infusion, within 2 hours prior to NTX-1088 administration, at a dose of 200 mg on Day 1 of every 21-day cycle.
  Interventions: Drug: NTX-1088; Drug: Pembrolizumab
- Part 2 - Dose Expansion (Monotherapy) (Experimental): NTX-1088 administered at the RP2D as a 60-minute IV infusion as a monotherapy.
  Interventions: Drug: NTX-1088
- Part 2 - Dose Expansion (Combination Therapy) (Experimental): NTX-1088 administered at the RP2D as a 60-minute IV infusion in combination with pembrolizumab at the standard labeled dose.
  Interventions: Drug: NTX-1088; Drug: Pembrolizumab

INTERVENTIONS:
Drug: NTX-1088 — IgG4 mAb targeting the poliovirus receptor (PVR, CD155).
Drug: Pembrolizumab — IgG4 mAb with high specificity of binding to the PD-1 receptor, thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2).
  Other Names: KEYTRUDA®
  Arms: Part 1 - Dose Escalation Phase (Combination Therapy); Part 2 - Dose Expansion (Combination Therapy)

SUMMARY:
This is a Phase 1,open-label, multi-center, first-in-human, 2-part (Part 1: dose escalation and Part 2: expansion) study, evaluating multiple doses and schedules of intravenously (IV) administered NTX-1088, with or without pembrolizumab, in patients with advanced solid malignancies (i.e., locally advanced or metastatic).

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multi-center study whose principal Part 1 stage objective is to determine the recommended Phase 2 dose (RP2D) of the anti-PVR monoclonal antibody (mAb) as a single agent and combined with the anti-PD-1 mAb pembrolizumab in patients with advanced solid malignancies.

In the Part 2 stage, the antitumor activity of NTX-1088 alone or combined with pembrolizumab will be evaluated in patients with malignancies known to express PVR.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have histologic or cytologic evidence of an advanced (locally advanced or metastatic) malignant solid cancer known to express PVR, including colorectal carcinoma (MSI-H and MSS with no liver mets), hepatocellular carcinoma, gastric/gastroesophageal junction/esophageal carcinoma, Non-Small Cell Lung Cancer (NSCLC), endometrial carcinoma, cervical carcinoma, Squamous Cell Carcinoma of the Head and Neck (SCCHN), Renal Cell Carcinoma (RCC), cutaneous melanoma, Basal Cell Carcinoma (BCC) or another tumor type approved by the Medical Monitor.
2. Except for dose escalation with pembrolizumab for patients in whom mAbs targeting PD-1 as monotherapy are the standard of care, patients enrolled in the dose-escalation parts must have disease that is resistant to or relapsed following available standard systemic therapy, or for which there is no standard systemic therapy or reasonable therapy in the physician's judgment likely to result in clinical benefit, or if such therapy has been refused by the patient. Documentation of the reason must be provided for patients who have not received a standard therapy likely to result in clinical benefit.
3. Patient must have received no more than 4 prior systemic therapies. Special cases of >4 prior systemic therapies will be discussed between the investigator and the Sponsor's medical team.
4. A fresh tumor biopsy will be required if the biopsy procedure is not a significant risk procedure defined as one without mortality or major morbidity in the patient's clinical setting and at the institution completing the procedure is estimated to be ≥2%. The Medical Monitor must be contacted to review documentation of biopsy risk.

   1. Patients enrolled in the dose-escalation part at relevant NTX-1088 doses (i.e., NTX-1088 at a dose >400 mg) will be required to undergo a tumor biopsy during the screening period and at the end of Cycle 2 (±7 days from C3D1), if the procedure is not a significant risk procedure as defined above.
   2. Patients enrolled in the expansion part will be required to undergo a tumor biopsy during the screening period and at the end of Cycle 2 (±7 days from C3D1), if the procedure is not a significant risk procedure as defined above.
5. The patient must have disease that is measurable by RECIST, version 1.1 (APPENDIX A) as assessed by the local site Investigator/radiology. For patients with prior radiation therapy, measurable lesions must be outside of any prior radiation field(s), unless disease progression has been documented at that site after radiation.
6. The patient is ≥18 years old on the day of signing the consent form.
7. The patient has an ECOG PS of ≤1.
8. The patient has life expectancy of >3 months
9. The patient has adequate baseline organ function, as demonstrated by the following:

   a. CrCL ≥30 mL/min as calculated by the Cockcroft-Gault formula: i. CrCl (male) = ([140-age] × weight in kg)/ (serum creatinine ×72) ii. CrCl (female) = CrCl (male)×0.85 b. Bilirubin ≤1.5×ULN. c. AST and ALT ≤2.5×ULN. Patients may have ALT and AST <5×ULN if the patient has hepatic metastases.

   d. Corrected calcium <11g/dL e. Albumin >3g/dL
10. For patients not taking warfarin or other oral anticoagulants: international normalized ratio (INR) ≤1.5 or prothrombin time (PT) ≤1.5×ULN; and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) ≤1.5×ULN. Patients taking warfarin should be on a stable dose that results in a stable INR <3.5. Among patients receiving other oral anticoagulant therapy, PT or aPTT must be within the intended therapeutic range of the anticoagulant and/or subcutaneous therapies should be monitored as standard per institution.
11. The patient has adequate baseline hematologic function, as demonstrated by the following:

    1. ANC ≥1.5×109/L.
    2. Hemoglobin ≥9 g/dL and no red blood cell transfusions during the prior 14 days.
    3. Platelet count ≥100×109/L and no platelet transfusions during the prior 14 days.
12. The patient has a left ventricular ejection fraction (LVEF) ≥45% as determined by either echocardiography (ECHO) or multigated acquisition (MUGA) scanning.
13. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Documented to be surgically sterile or postmenopausal (amenorrhea 24 months and follicle-stimulating hormone [FSH] ≥30 mIU/mL), OR
    2. Practicing true abstinence for at least 28 days prior to study treatment until 120 days after the last dose of study treatment and having a negative serum or urine pregnancy test within 72 hours before initiating treatment, or in closer proximity to treatment start-date as required by local/institutional regulations, OR
    3. Using 2 forms of highly effective contraception, including 1 physical barrier (condom or diaphragm) plus another method, such as adequate hormonal method (e.g., contraceptive implants, injectables, oral contraceptives) or nonhormonal methods (e.g., intrauterine device, spermicidals) from screening or at least 28 days prior to study treatment administration (whichever is earlier) until 120 days after the last dose of study treatment and having a negative serum or urine pregnancy test within 72 hours before initiating treatment, or in closer proximity to treatment start-date as required by local/institutional regulations.
14. Male patients with female partners of childbearing potential may be enrolled if they are:

    1. Documented to be surgically sterile (vasectomy), OR
    2. Practicing true abstinence until 120 days after the last dose of study treatment, OR
    3. Using 2 effective methods of contraception including one barrier method (e.g., condom with spermicide and contraception by female partner) for the duration of time on the study and for 3 months after administration of the last dose of study treatment, unless their partners are infertile or surgically sterile.
15. The patient has signed the Informed Consent Form (ICF) prior to initiation of any study-specific procedures or treatment.
16. The patient can adhere to the study visit schedule and other protocol requirements, including follow-up for survival assessment.
17. The patient has sufficient venous access enabling plasma/blood sampling as per protocol.

Exclusion Criteria:

1. The patient (for combination arm only) was discontinued from treatment with an immuno-oncology therapeutic due to a Grade 3 or higher immune-related adverse event (irAE) except endocrine disorders that can be treated with replacement therapy or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis. This does not apply to irAEs due to prior treatment with cell therapy.
2. The patient has received prior radiotherapy within 2 weeks of treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation with a limited port ≤2 weeks of radiotherapy to non-central nervous system (CNS) disease.
3. The patient has received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of study medication.
4. The patient has received treatment with approved anticancer therapies including cytotoxic chemotherapy, monoclonal antibodies, and/or small molecule tyrosine kinase inhibitors within 14 days prior to study therapy administration or 5 half-lives, whichever is shorter (42 days for nitrosourea or mitomycin-C); patients with advanced prostate cancer who are receiving luteinizing hormone releasing hormone (LHRH) agonists are permitted onto the study and should continue use of these agents during study treatment.
5. The patient has had an allogeneic tissue/solid organ transplant.
6. The patient has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention.
7. The patient has received prior treatment with another investigational agent that targets PVR.
8. If the patient had major surgery, the patient must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
9. The patient is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks or 5 half-lives, whichever is shorter, prior to the first dose of study treatment.
10. The patient must have recovered from all AEs due to previous therapies to Grade ≤1 or baseline. Patients with Grade ≤2 alopecia and/or neuropathy may be eligible. Patients with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible. Prior toxicities that resulted in laboratory abnormalities should have resolved to Grade ≤1 unless a higher-grade abnormality is allowed by the inclusion criteria. If medical therapy is required for the treatment of a laboratory abnormality, the dose and laboratory value(s) should be stable.
11. The patient has an active autoimmune disease that required systemic treatment in the past. Patients who have not required systemic treatment for at least two years may be enrolled if permission is provided after discussion with the Medical Monitor (replacement therapy, e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a form of systemic treatment, and is allowed).
12. The patient has an uncontrolled endocrine disorder.
13. The patient has clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association Class 3 or 4 heart failure [see Section 8.2.7]), uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension, or clinically significant arrhythmias not controlled by medication).
14. The patient has a history of (non-infectious) pneumonitis or interstitial pulmonary disease that required steroids or has current pneumonitis or interstitial pulmonary disease.
15. The patient has uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study.
16. The patient has had a severe hypersensitivity reaction (Grade ≥3) to pembrolizumab and/or any of its excipients (pembrolizumab combination enrollment only).
17. The patient has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
18. The patient has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection requiring therapy, disseminated intravascular coagulation, psychiatric illness, drug abuse, or a social situation that would limit compliance with study requirements.
19. The patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
20. The patient has known positive status for human immunodeficiency virus (HIV). No HIV testing is required unless mandated by local health authority.
21. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen reactive) or known active Hepatitis C virus (defined as HCV RNA detected) infection. Testing for Hepatitis B and Hepatitis C is not required unless mandated by a local health authority.
22. The patient is oxygen dependent.
23. The patient has any medical condition which, in the opinion of the Investigator, places the patient at an unacceptably high risk for toxicities.
24. The patient has an additional active malignancy that is progressing or has required active treatment within the past 3 years. Patients with a past cancer history with substantial potential for recurrence must be discussed with the Medical Monitor before study entry. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including transitional cell carcinoma, cervical intraepithelial neoplasia, breast cancer, and melanoma in situ), organ-confined prostate cancer with no evidence of PD.
25. The patient has known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging, clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment. For patients with a history of CNS involvement, the repeat imaging should be performed during study screening. However, CNS imaging is not required prior to study entry unless there is clinical suspicion of CNS involvement.
26. The patient is pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | First 21 days of treatment.
  The incidence of DLTs during the DLT assessment period.
Dose-Finding | Screening to 30 days from last dose.
  Determination of the MTD or maximum tested dose, and the RP2D.
Frequency and Severity of Adverse Events (AE) | Screening to 30 days from last dose.
  The incidences and percentages of patients experiencing AEs summarized by NCI CTCAE version 5.0 grade and by causality.

SECONDARY OUTCOMES:
Pharmacokinetics of NTX-1088 | Day 1 of dosing through 21 days post last dose.
  Maximum Plasma Concentration (Cmax)
Pharmacokinetics of NTX-1088 | Day 1 of dosing through 21 days post last dose.
  Area Under the Curve (AUC)
Objective Response Rate (ORR) | Day 1 of dosing through 90 days after the last dose.
  ORR according to RECIST v1.1.
Duration of Response (DoR) | Day 1 of dosing through 90 days after the last dose.
  Time from the date measurement criteria are first met for PR or CR to the date measurement criteria are first met for progressive disease.
Progression Free Survival (PFS) | Day 1 of dosing through 90 days after the last dose.
  Time from the date of initiation of study therapy to the date measurement criteria are first met for progressive disease or death from any cause, whichever occurs first.
Overall Survival (OS) | Day 1 of dosing through 90 days after the last dose.
  Time from the date of initiation of study therapy to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - City of Hope, Duarte, California
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Maria Skłodowska-Curie National Research Institute of Oncology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No